CLINICAL TRIAL: NCT04768270
Title: Drug Screening of Patient-derived Organoids From Ovarian Cancer Culture to Personalized Therapy,an Exploratory Research
Brief Title: The Culture of Ovarian Cancer Organoids and Drug Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Other Study IDs: CQGOG0201
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer
Keywords: tumor organoids; drug sensitivity; precision treatment
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Ovarian cancer tissues were cut into 1-3 mm3 pieces. Two random pieces were snap frozen and stored at -80℃ for DNA isolation, two random pieces were fixed in formalin for histopathological analysis, and the remainder was processed for organoids.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — It is an observation trial.

SUMMARY:
The tumor organoids platform can provide the precise genetic information and phenotype, as well as the heterogeneity of the tumor, thus provide information on drug sensitivity specific to the patient.This is an exploratory research to see if organoids testing could help guide precision treatment for ovarian cancer(OC) patients.

DETAILED DESCRIPTION:
Tissue will be received from operative specimens( primary ovarian carcinoma) at time of primary cytoreductive surgery.Ovarian cancer(OC) organoids will be then cultured. Organoids will be validated with a combination of Next Generation Sequencing (NGS) analysis and immunohistochemistry (TP53, PAX8 etc). After then, the patient-derived organoids cultured from OC will be compared the sensitivity to standard regimens (chemotherapies and targeted agents) recommendated by NCCN guidlines versus patients treated in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Ovarian cancer patients who will accept primary cytoreductive surgery, with histopathological type: low/high grade serous carcinoma, clear cell carcinoma, endometrioid carcinoma, mucinous carcinoma.
2. ECOG score 0~1,age 18~70 years old
3. Expected survival over 6 months
4. The serum or urine pregnancy test must be negative within 7 days before enrollment for the women of childbearing age who should agree that contraception must be used during the trial
5. CBC：Hb≥70g/L、WBC≥3.5×109/ L 、ANC≥1.5×109/L、PLT≥80×109/L；
6. Serum ALT≤2×UL, AST≤2×ULN；Serum creatinine≤1.5×ULN；

Exclusion Criteria:

1. Activity or uncontrol severe infection
2. Liver cirrhosis, Decompensated liver disease
3. History of immune deficiency, including HIV positive or suffering from congenital immunodeficiency disease
4. Chronic renal insufficiency or renal failure
5. Has combined with other malignant tumor which diagnosed within 5 years and/or needed to be treated
6. Myocardial infarction, severe arrhythmia and NYHA (New York heart association)≥2 for congestive heart failure
7. During the treatment for complications, the drugs which lead to serious liver and/or kidney function impairment need to be used, such as tuberculosis

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: ovarian cancer patients who accept primary cytoreductive surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  Progression-free survival
OS | 5 years
  Overall survival

SECONDARY OUTCOMES:
ORR | 1 year
  CR+PR
DCR | 1 year
  CR+PR+SD

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China